CLINICAL TRIAL: NCT04489979
Title: Analgetics vs Analgetics and Antibiotics for Pediatric Clinical and Sonographic Orchitis or Epididymitis
Status: Completed | Type: Observational
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Principal Investigator, Erez Nadir, MD, Neonatologist, Hillel Yaffe Medical Center
Other Study IDs: 0012-20-HYMC
Record Dates: First submitted 2020-02-29; First posted 2020-07-28 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Epididymitis Orchitis
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Analgetics only: Children with epididymitis / orchitis treated by analgetics only.
  Interventions: Other: Antibiotics
- Analgetics and antibiotics: Children with epididymitis / orchitis treated by analgetics and antibiotics.
  Interventions: Other: Antibiotics

INTERVENTIONS:
Other: Antibiotics — Children with epididymitis / orchitis who were treated by antibiotics in addition to analgetics.

SUMMARY:
Some children are admitted to pediatric emergency department due to epididymitis or orchitis. Some of them are treated by analgetics only whie some are treated by analgetics with antibiotics. The study will compare clinical presentation between groups and will compare pediatric urologic outpatient clinic follow up findings.

DETAILED DESCRIPTION:
Some children are admitted to pediatric emergency department due to epididymitis or orchitis. Some of them are treated by analgetics only whie some are treated by analgetics with antibiotics. The study will compare clinical presentation between groups and will compare pediatric urologic outpatient clinic follow up findings.

ELIGIBILITY:
Inclusion Criteria:

* All children admitted to pediatric emergency department due to epididymitis or orchitis

Exclusion Criteria:

* No sonographic or laboratory exam
* Antibiotic treatment before diagnosis
* No outpatient follow-up
* Known urologic congenital malformations
* Admission to inpatient department or emergency surgery

Max Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Only males have testicles
Study Population: Male children who were admitten to pediatric emergency department due to epididymitis or orchitis
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Healing | 1 month
  No symptoms any more

CONTACTS AND LOCATIONS:
Overall Officials: Erez Nadir, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe medical center, Hadera, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lau P, Anderson PA, Giacomantonio JM, Schwarz RD. Acute epididymitis in boys: are antibiotics indicated? Br J Urol. 1997 May;79(5):797-800. doi: 10.1046/j.1464-410x.1997.00129.x. PMID 9158522